CLINICAL TRIAL: NCT00337467
Title: Phase IIIb Multicenter, Single Arm, Open-Label Pilot Study to Evaluate the Effectiveness and Safety of Maintenance With Atazanavir/Ritonavir as Single Enhanced Protease Inhibitor Therapy in HIV-Infected Patients Evidencing Virologic Suppression OREY (Only REYataz) Study
Brief Title: Phase IIIb Study to Evaluate the Effectiveness and Safety of Atazanavir/Ritonavir as Single Enhanced Protease Inhibitor Therapy in Human Immunodeficiency Virus (HIV)-Infected Subjects Evidencing Virologic Suppression
Acronym: OREY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-227
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-06

CONDITIONS: Human Immunodeficiency Virus (HIV) Infections
Keywords: HIV-Infected Patients Evidencing Virologic Suppression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — atazanavir, ritonavir drug combination; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Atazanavir + Ritonavir

INTERVENTIONS:
Drug: Atazanavir + Ritonavir — Capsules, Oral, ATV 300mg + RTV 100mg, once daily, 96 weeks
  Other Names: Reyataz; BMS-232632

SUMMARY:
The main purpose is to explore whether atazanavir/ritonavir (ATV/RTV) single enhanced protease inhibitor therapy can maintain virologic suppression without a marked increase in virologic failure.

ELIGIBILITY:
Inclusion Criteria:

* On continued antiretroviral (ARV) treatment, with no discontinuation periods, for the previous 6 months (24 weeks).
* Absence of evidence or suspected virologic failure on antiretroviral therapy
* Absence of known primary mutations in the protease gene
* Only 1 highly active antiretroviral therapy (HAART) prior to current one
* HIV RNA < 50 copies/mL in the last 6 months (single blip below 200 c/mL allowed)
* On ATV/RTV +2 nucleoside reverse transcriptase inhibitors (NRTIs) (or 1 NRTI + tenofovir [TDF]) for at least 8 weeks before study entry, without treatment-limiting adverse effects

Exclusion Criteria:

* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment.
* Active disease condition (e.g. moderate to severe hepatic impairment/active renal disease/history of clinically significant heart conduction disease)
* Patients with chronic hepatitis B receiving lamivudine (3TC), Tenofovir Disoproxil Fumarate (TDF) or emtricitabine (FTC).
* CD4 < 100 cells/mm3
* Grade IV laboratory values: Hemoglobin < 6.5 g/dL or white blood cells (WBC) <800/mmm3 or absolute neutrophil count < 500/mm3, or platelets < 20,000/mm3 or diffuse petechiae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Spain (3):
  - Local Institution, Córdoba
  - Local Institution, Madrid
  - Local Institution, Málaga

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 63 participants were enrolled in this study; 2 were never treated (1 no longer met study criteria and 1 concomitant medication not permitted).
Groups:
- Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.: ATV/RTV treatment regimen was administered once daily. ATV: 2 x 150 mg capsules once daily with food (meal or snack), RTV: 1 x 100 mg capsule once daily with food (meal or snack)
Period: Overall Study
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Started | 61
Discontinued Prior to Week 96 | 10 (5 of these participants discontinued prior to Week 48)
Completed | 51
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Subject Withdrew Consent | 2
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 2
Not completed — Subject No Longer Met Study Criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 46
Race/Ethnicity, Customized [Number; unit: participants]
  White | 61
Cluster of Differentiation 4 (CD4) Categories [Number; unit: participants]
  CD4 Count <200 cells/mm3 | 3
  CD4 Count >=200 cells/mm3 | 58
Human Immunodeficiency Ribonucleic Acid (HIV RNA) Categories [Number; unit: Participants]
  HIV RNA <50 c/mL | 60
  HIV RNA >=50 c/mL | 1
CD4 Count [Mean (Standard Deviation); unit: cell/mm3] | 559 (272.8)
Fasting High-Density Lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population analyzed = 54 (treated participants with baseline measure)
  mg/dL | 45 (10.4)
Fasting Low-Density Lipoprotein (LDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population analyzed = 54 (treated participants with baseline measure)
  mg/dL | 112 (52.3)
Fasting Non-HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population analyzed = 54 (treated participants with baseline measure)
  mg/dL | 144 (57.9)
Fasting Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population analyzed = 54 (treated participants with baseline measure)
  mg/dL | 189 (57)
Fasting Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Population analyzed = 54 (treated participants with baseline measure)
  mg/dL | 164 (95.7)
HIV RNA [Mean (Standard Deviation); unit: log10 c/mL] | 1.71 (0.152)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Failure Through Week 48
Description: Treatment Failure through Week 48 defined as virologic rebound (HIV RNA >=400 c/mL) on or before Week 48 or study discontinuation before Week 48. Virological rebound is defined as confirmed on-treatment HIV ribonucleic acid (RNA) >= 400 c/mL at 2 consecutive visits or last on-treatment HIV RNA >=400 c/mL followed by discontinuation of study therapy.
Time Frame: Week 48
Population: Treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy
Number analyzed (Participants) | 61
Percentage of Participants | 21.3
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Test type: Superiority or Other; exact binomial methods; Given the small sample size, the 95% confidence interval is made with exact binomial methods; Percentage of Participants = 21.3, 95% CI 2-sided [11.9 to 33.7]

2. Secondary Outcome: Percentage of Participants With Treatment Failure Through Week 96
Description: Treatment Failure through Week 96 defined as virologic rebound (HIV RNA >=400 c/mL) on or before Week 96 or study discontinuation before Week 96. In addition, treatment failure defined based on HIV RNA >= 50 c/mL, latter analysis performed on treated subjects with baseline HIV RNA < 50 c/mL.
Time Frame: Week 96
Population: Treated participants. For the second row (n=60), one subject was excluded because of baseline HIV RNA > 50 c/mL.
Measure: Number; unit: percentage of participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy
Number analyzed (Participants) | 61
percentage of participants
  HIV RNA >= 400 c/mL(n=61) | 34.4
  HIV RNA>=50 c/mL w/Baseline HIV RNA<50 c/mL (n=60) | 43.3
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Test type: Superiority or Other; exact binomial methods; Given the small sample size, the 95% confidence interval is made with exact binomial methods; Percentage of Participants = 34.4, 95% CI 2-sided [22.7 to 47.7]

3. Secondary Outcome: Percentage of Participants With Virological Rebound Through Week 48
Description: Virological rebound is defined as confirmed on-treatment HIV RNA >= 400 c/mL at 2 consecutive visits or last on-treatment HIV RNA >=400 c/mL followed by discontinuation of study therapy. In addition, virologic rebound defined based on HIV RNA >=50 c/m, latter analysis performed on subjects with baseline HIV RNA < 50 c/mL.
Time Frame: Week 48
Population: Treated participants. For the second row (n=60), one subject was excluded because of baseline HIV RNA > 50 c/mL.
Measure: Number; unit: percentage of participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy
Number analyzed (Participants) | 61
percentage of participants
  HIV RNA >= 400 c/mL (n=61) | 12
  HIV RNA>=50 c/mL w/Baseline HIV RNA<50 c/mL (n=60) | 26.7

4. Secondary Outcome: Percentage of Participants With Virological Rebound Through Week 96
Description: as for outcome 3
Time Frame: Week 96
Population: Treated participants. For the second row (n=60), one subject was excluded because of baseline HIV RNA > 50 c/mL.
Measure: Number; unit: percentage of participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy
Number analyzed (Participants) | 61
percentage of participants
  HIV RNA >= 400 c/mL (n=61) | 14.8
  HIV RNA>=50 c/mL w/Baseline HIV RNA<50 c/mL (n=60) | 33.3

5. Secondary Outcome: Cumulative Proportion of Participants Without Treatment Failure Through Week 100
Description: This Kaplan-Meier life table reports the cumulative proportion of participants without treatment failure up to the end of the respective time interval. Failure time is measured from the start of study therapy, and is based on the earliest event defining failure (virologic rebound at or before Week 96, or discontinuation prior to Week 96).
Time Frame: Through Week 100
Population: treated participants; n= the number at risk entering interval
Measure: Number; unit: proportion of participants
Groups:
- Proportion of Participants: Proportion of participants without treatment failure at the end of interval
Arm/Group | Proportion of Participants
Number analyzed (Participants) | 61
proportion of participants
  Interval Week 4 - 8 (n=61) | 0.9836
  Interval Week 8 - 12 (n=60) | 0.9508
  Interval Week 12 - 16 (n=58) | 0.9016
  Interval Week 16 - 20 (n=55) | 0.8852
  Interval Week 20 - 24 (n=54) | 0.8689
  Interval Week 24 - 28 (n=53) | 0.8525
  Interval Week 32 - 36 (n=52) | 0.8197
  Interval Week 36 - 40 (n=50) | 0.7869
  Interval Week 48 - 52 (n=48) | 0.7541
  Interval Week 56 - 60 (n=46) | 0.7377
  Interval Week 64 - 68 (n=45) | 0.7049
  Interval Week 68 - 72 (n=43) | 0.6885
  Interval Week 72 - 76 (n=42) | 0.6721
  Interval Week 84 - 88 (n=41) | 0.6557
  Interval Week 92 - 96 (n=40) | 0.6557
  Interval Week 96 - 100 (n=31) | 0.6557

6. Secondary Outcome: Proportion of Participants With Virologic Rebound Through Week 96
Description: Virologic rebound is defined as confirmed on-study HIV RNA ≥ 400 c/mL or last on-study HIV RNA ≥ 400 c/mL followed by treatment discontinuation.
Time Frame: Through Week 96
Population: This analysis was not done; however, percentage of participants with virologic rebound through Weeks 48 and 96 are reported in Secondary Outcome Measures 3 and 4. Time to reatment failure (defined as the earlier of virologic rebound or treatment discontinuation) is reported in Secondary Outcome Measure 5.
Measure: Number; unit: proportion of participants
Groups:
- Proportion of Participants: Proportion of participants without virologic rebound at the end of interval
Arm/Group | Proportion of Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: n=number of participants with CD4 cell count at baseline and at Week 24
Measure: Mean (Standard Deviation); unit: cells /mm3
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
cells /mm3
  Baseline Value (n=61) | 559 (272.8)
  Change at Week 24 (n=51) | 61 (173.3)
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change (Final Values) = 61, 95% CI 2-sided [12.3 to 109.8], Standard Error of Mean 24.3

8. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: n=number of participants with CD4 cell count at baseline and at Week 48.
Measure: Mean (Standard Deviation); unit: cells /mm3
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
cells /mm3
  Baseline Value (n=61) | 559 (272.8)
  Change at Week 48 (n=46) | 53 (203.5)
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change (Final Values) = 53, 95% CI 2-sided [-7.1 to 113.7], Standard Error of Mean 30.0

9. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: n=number of participants with CD4 cell count at baseline and at Week 96.
Measure: Mean (Standard Deviation); unit: cells /mm3
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
cells /mm3
  Baseline Value (n=61) | 559 (272.8)
  Change at Week 96 (n=40) | 63 (208.1)
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change (Final Values) = 63, 95% CI 2-sided [-4.0 to 129.1], Standard Error of Mean 32.9

10. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to AEs
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition that does not necessarily have a causal relationship to treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. AE grades are: mild (1), moderate (2), severe (3), life-threatening (4), and death (5).
Time Frame: From Baseline through Week 96
Population: Treated Participants
Measure: Number; unit: percentage of participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
percentage of participants
  All Grades AEs | 75.4
  All Grades AEs Related to Study Therapy | 13.1
  Grade 3 to Grade 4 AEs | 18
  Grade 3 to Grade 4 AEs Related to Study Therapy | 3.3
  Deaths | 3.3
  SAEs | 19.7
  SAEs Related to Study Therapy | 0
  AEs Leading to Discontinuation | 4.9
  Lipodystrophy-Related AEs | 1.6

11. Secondary Outcome: Mean Percent Changes From Baseline in Fasting Total Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Non-HDL Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, and Triglycerides at Week 48
Description: Lipid values after starting lipid-reducing agents are excluded from analyses. Baseline values are provided in Baseline Characteristics.
Time Frame: Baseline, Week 48
Population: n= number of treated participants with baseline measure and measure at Week 48
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
percent change
  Total Cholesterol (n=36) | 9 (18.0)
  HDL Cholesterol (n=35) | 2 (18.5)
  Non-HDL Cholesterol (n=35) | 12 (24.4)
  LDL Cholesterol (n=33) | 20 (33.4)
  Triglycerides (n=36) | 17 (51.4)
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Total Cholesterol at Week 48; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 9, 95% CI 2-sided [2.5 to 14.6], Standard Error of Mean 3.0
Statistical Analysis 2: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting HDL Cholesterol at Week 48; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 2, 95% CI 2-sided [-3.9 to 8.8], Standard Error of Mean 3.1
Statistical Analysis 3: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Non-HDL Cholesterol at Week 48; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 12, 95% CI 2-sided [4.0 to 20.8], Standard Error of Mean 4.1
Statistical Analysis 4: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting LDL Cholesterol at Week 48; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 20, 95% CI 2-sided [8.0 to 31.7], Standard Error of Mean 5.8
Statistical Analysis 5: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Triglycerides at Week 48; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 17, 95% CI 2-sided [-0.4 to 34.4], Standard Error of Mean 8.6

12. Secondary Outcome: Mean Percent Changes From Baseline in Fasting Total Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Non-HDL Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, and Triglycerides at Week 96
Description: as for outcome 11
Time Frame: Baseline, Week 96
Population: n=number of treated participants with baseline measure and measure at Week 96
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 61
percent change
  Total Cholesterol (n=29) | 14 (17.4)
  HDL Cholesterol (n=29) | 2 (21.2)
  Non-HDL Cholesterol (n=29) | 19 (23.7)
  LDL Cholesterol (n=28) | 29 (34.4)
  Triglycerides (n=29) | 16 (67.2)
Statistical Analysis 1: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Total Cholesterol at Week 96; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 14, 95% CI [6.9 to 20.1], Standard Error of Mean 3.2
Statistical Analysis 2: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting HDL Cholesterol at Week 96; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 2, 95% CI 2-sided [-6.0 to 10.2], Standard Error of Mean 3.9
Statistical Analysis 3: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Non-HDL Cholesterol at Week 96; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 19, 95% CI 2-sided [10.3 to 28.4], Standard Error of Mean 4.4
Statistical Analysis 4: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting LDL Cholesterol at Week 96; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 29, 95% CI 2-sided [15.3 to 42.0], Standard Error of Mean 6.5
Statistical Analysis 5: Comparison: Atazanavir (ATV)/Ritonavir (RTV) Monotherapy; Percent Change from Baseline in Fasting Triglycerides at Week 96; Test type: Superiority or Other; normal approximation for 95% CI; Mean Change = 16, 95% CI 2-sided [-9.5 to 41.6], Standard Error of Mean 12.5

13. Secondary Outcome: Number of Participants With Genotype Substitutions for Virologic Rebounds (HIV-RNA ≥ 400 c/mL) Through Week 48
Description: International Aids Society of the United States (IAS-USA)-defined major protease inhibitor (PI) substitutions are V32I, L33F, M46I/L, I47V, G48V, I50L/V, I54M/L, I76V, I82A/F/T/S, I84V, N88S, and L90M. Reverse Transcriptase (RT) are TAMS and M184V.
Time Frame: Week 48
Population: Number of participants with virologic rebounds (HIV-RNA ≥ 400 c/mL) through Week 48.
Measure: Number; unit: participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy.
Number analyzed (Participants) | 7
participants
  IAS-USA-defined major PI substitutions | 1
  RT substitutions | 0

14. Secondary Outcome: Number of Participants With Genotype Substitutions for Virologic Rebounds (HIV-RNA ≥ 400 c/mL) Through Week 96
Description: as for outcome 13
Time Frame: Week 96
Population: Number of participants with virologic rebounds (HIV-RNA ≥ 400 c/mL) through Week 96.
Measure: Number; unit: participants
Arm/Group | Atazanavir (ATV)/Ritonavir (RTV) Monotherapy
Number analyzed (Participants) | 9
participants
  IAS-USA-defined major PI substitutions | 2
  RT substitutions | 0

ADVERSE EVENTS:
Groups:
- ATV/RTV Monotherapy: ATV/RTV treatment regimen was administered once daily. ATV: 2 x 150 mg capsules once daily with food (meal or snack), RTV: 1 x 100 mg capsule once daily with food (meal or snack)
Arm/Group | ATV/RTV Monotherapy
Serious Adverse Events (participants affected / at risk) | 12/61
Other Adverse Events (participants affected / at risk) | 25/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV Monotherapy (N=61)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1
DYSTHYMIC DISORDER (Psychiatric disorders) | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 1
DEPRESSION SUICIDAL (Psychiatric disorders) | 1
HEADACHE (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
SEPSIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
APPENDICITIS (Infections and infestations) | 1
EYE INFECTION SYPHILITIC (Infections and infestations) | 1
TESTICULAR ATROPHY (Reproductive system and breast disorders) | 1
ACCIDENT (Injury, poisoning and procedural complications) | 1
MULTI-ORGAN FAILURE (General disorders) | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV Monotherapy (N=61)
DEPRESSION (Psychiatric disorders) | 4
HEADACHE (Nervous system disorders) | 5
TOOTH INFECTION (Infections and infestations) | 4
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 7
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.